CLINICAL TRIAL: NCT07134738
Title: Multicenter, Open-label, Non-interventional Study to Assess the Safety and Tolerability of Dimolegin® as a Means of Preventing Thrombotic Complications in the Complex Therapy of Hospitalized Patients With Moderate COVID-19 in a Real Clinical Practice
Brief Title: Dimolegin® (60 mg) for Patients With Moderate COVID-19: A Non-Interventional Study
Status: Completed | Type: Observational
Sponsor: Avexima Diol LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AVD-DIM-PM-2023-15
Record Dates: First submitted 2025-08-08; First posted 2025-08-21 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — (+-)-(1'R*,2'S*,6'R*)-(2-hydroxy-4,6-dimethoxyphenyl)(3'-methyl-2'-(3''-methylbut-2''-enyl)-6-phenylcyclohex-3'-enyl)methanone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1 (Dimolegin® Group): Dimolegin® is administered orally once dailyюThe recommended dose is 60 mg once daily. Treatment duration depends on clinical indication and may last up to 30 days.
  Interventions: Drug: Dimolegin

INTERVENTIONS:
Drug: Dimolegin — Dimolegin® is administered orally once daily,The recommended dose is 60 mg (six 10 mg tablets) once daily.

SUMMARY:
A multicenter, open-label, non-interventional study evaluates the safety and tolerability of oral Dimolegin® (60 mg once daily) for thromboprophylaxis in hospitalized adults (≥18 years) with moderate COVID-19 in real clinical pratice. The primary objective is to assess safety and tolerability of Dimolegin® in preventing thrombotic complications.

ELIGIBILITY:
Inclusion Criteria:

Here's a concise English translation:

* Voluntarily signed informed consent to participate in a non-interventional study.
* Hospitalized patients with moderate COVID-19 requiring anticoagulant therapy for prevention of thrombotic complications.
* Men and women aged ≥18 years.
* Patients prescribed Dimolegin® 10 mg enteric-coated film tablets for thromboprophylaxis as part of routine care for moderate COVID-19.
* Ability to understand study requirements, provide written consent and comply with protocol procedures.

Exclusion Criteria:

* Hypersensitivity to Dimolegin®.
* Clinically significant active bleeding at screening.
* Concomitant therapy with fibrinolytics or other anticoagulants.
* Anemia or thrombocytopenia.
* Thrombophilia.
* Other coagulopathies or contraindications to anticoagulants.
* Liver disease with impaired function or biliary tract disease.
* Creatinine clearance <30 mL/min.
* Gastrointestinal disorders affecting absorption.
* Pregnancy, breastfeeding, suspected pregnancy, or planned pregnancy within 3 months (including male patients whose partners plan pregnancy).
* Use of investigational or unapproved drugs, or participation in another clinical study within 90 days before therapy start.
* History or suspicion of alcohol or drug abuse, dependence, or addiction.
* Any other condition that, in the investigator's opinion, could interfere with study participation or pose undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized adult patients (≥18 years) with moderate COVID-19 requiring thromboprophylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Frequency of major bleeding events | through discharge from the hospital, up to 30 days

SECONDARY OUTCOMES:
Frequency of major bleeding events | up to 60±3 days
Frequency of moderate bleeding events | up to 60±3 days
Frequency of minor bleeding events | up to 60±3 days
Frequency of anemia | up to 60±3 days
Frequency of AR of special interest regardless of severity | up to 60±3 days
Proportion of patients with ARs and SARs | up to 60±3 days
Change from baseline in INR, APTT, prothrombin time, and D-dimer levels | through discharge from the hospital, up to 30 days
Frequency of gastrointestinal symptoms | through discharge from the hospital, up to 30 days

CONTACTS AND LOCATIONS:
Locations (6):
- Russia (6):
  - Regional Clinical Hospital No. 3, Chelyabinsk
  - Republican Clinical Hospital named after Professor A.F. Agafonov, Kazan'
  - Infectious Diseases Clinical Hospital No. 1, Moscow
  - Infectious Diseases Hospital No. 2, Sochi
  - Tomsk Regional Hospital, Tomsk
  - Regional Infectious Diseases Clinical Hospital, Yaroslavl

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chulanov V, Sagalova O, Khaertynov H, Teteneva A, Kravchenko I, Balashov O, Makarov D, Sychev D. Safety of a Domestic Original Direct Oral Anticoagulant from the Group of Factor Xa Inhibitors in the Prevention of Thrombotic Complications in Patients with COVID-19 in Real Clinical Practice. Clinical infectology and parasitology. 2025, 14 (3): 347-361. (In Russ.) DOI: 10.34883/PI.2025.14.3.038